CLINICAL TRIAL: NCT04708795
Title: Clinical Trial on Pharmacokinetic and Tolerability of AP701
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CannaXan GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SELECT
Record Dates: First submitted 2020-12-21; First posted 2021-01-14 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetic; Tolerability; Safety
Keywords: Cannabis; Cannabis based medicine; THC; Tetrahydrocannbinol
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verum (Experimental): AP701 single dose oromucosal application
  Interventions: Drug: AP701

INTERVENTIONS:
Drug: AP701 — Preparation of Cannabis flowers (Cannabis flos)

SUMMARY:
This study aims to investigate the uptake of AP701, a preparation from cannabis flowers, into the bloodstream after in single administration in healthy volunteers.

DETAILED DESCRIPTION:
Pharmacokinetic parameters and tolerability of AP701 is studied over 30 hours after single dose administration in healthy volunteers in a prospective and open-label manner at a single study center.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Male in the age of 35 - 60 year at study start
3. Body mass index of 18 to 30 kg/m2
4. Non-smoker, no use of any Tabaco products
5. Good general health status (Karnofsky Score = 100)
6. Current ECG without abnormal findings (i.a. QTcF < 450 ms)
7. Physical examination, medical history without exclusionary findings
8. Pulse rate between 50 and 90 bpm
9. Blood pressure between systolic 90 - 140 mmHg, diastolic 50 - 90 mmHg
10. Lab values for liver function (ALT, AST, AP, Bilirubin total) within normal ranges
11. Lab values for renal function (S-Creatinine, eGFR) within normal range
12. Negative test result on HIV I, HIV II, hepatitis B cell surface antigen, hepatitis C antibody
13. Negative test result of urine screening for Cannabis, alcohol, and substance abuse

Exclusion Criteria:

1. Medical history of hypersensitivity or intolerance to the investigational product or its ingredients or to ingredients of similar chemical structure
2. Use of Cannabis products within the last 8 weeks
3. Use of opioids
4. Former or present dependency (e.g. to alcohol, medicinal products, drugs)
5. Participation in another clinical trial within the last four weeks prior to study inclusion
6. Present, former, or family history of mental illnesses such as severe de pression, psychosis, bipolar disorder, mania, obsessive compulsive disorder, and anxiety disorder
7. Acute severe somatic disease (e.g. gastrointestinal diseases, influenza)
8. Body temperature ≥ 38 °C
9. Present cardiovascular, respiratory, diabetic, or cancer disease
10. Hepatitis or other liver and renal disease
11. Other diseases or conditions that do not allow the participant to assess the nature and scope, and possible consequences of participating in this clinical trial
12. Indications that the participant is unlikely to comply with the study protocol (e.g. lack of cooperation)
13. Taking any pharmaceutical products (including any medication interacting with metabolism of THC, e.g. St. John's wort)

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of pharmacokinetic parameter of THC (area under the curve) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of THC (maximum observed drug concentration) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of THC (time to reach maximum drug concentration) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of THC (area under the curve from timepoint zero to quantification limits) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to detection limits after application of investigational product
Evaluation of pharmacokinetic parameter of THC (area under the curve from 0 to 24 hours) | 24 hours
  Pharmacokinetic outcome of THC measured 0 to 24 hours after application of investigational product
Evaluation of pharmacokinetic parameter of THC (last drug concentration above quantification limits) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of THC (time of last drug concentration above quantification limits) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of THC (half-life associated with the terminal slope) | 30 hours
  Pharmacokinetic outcome of THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (area under the curve) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (maximum observed drug concentration) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (time to reach maximum drug concentration) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (area under the curve from timepoint zero to quantification limits) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (area under the curve from 0 to 24 hours) | 24 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 24 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (last drug concentration above quantification limits) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (time of last drug concentration above quantification limits) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Evaluation of pharmacokinetic parameter of 11-OH-THC (half-life associated with the terminal slope) | 30 hours
  Pharmacokinetic outcome of 11-OH-THC measured 0 to 30 hours after application of investigational product
Adverse events (AE) | 30 hours
  Number and severity of adverse events (AE)
Pschotropic drug effects measured by questionnaire | 30 hours
  Questionnaire comprising 17 questions on intoxication to be answered on numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lorenzl, PhD, Principal Investigator — Phase I Unit of CannaXan GmbH
Locations (1):
- Phase I Unit of CannaXan GmbH, Warngau, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No